CLINICAL TRIAL: NCT02088346
Title: Intravenous Thrombolysis Guided by Telemedicine Consultation System for Acute Ischemic Stroke Patients in China
Brief Title: Acute Stroke Advancing Program Using Telemedicine
Acronym: ASAP-Tel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Department of Science and Technology of Shanxi Province (Unknown); Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Other Study IDs: Xijing-Tele-001
Record Dates: First submitted 2014-02-27; First posted 2014-03-14 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2014-09

CONDITIONS: Stroke
Keywords: Stroke; Thrombolysis; Tissue plasminogen activator; Urokinase; Telemedicine
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Teleconsultation: Intravenous thrombolysis guided by telemedicine consultation system based on portable hardwares
  Interventions: Other: Telemedicine consultation system
- Historical control: Usual stroke care without the guidance from hub hospital

INTERVENTIONS:
Other: Telemedicine consultation system — Telemedicine consultation system based on portable hardwares
  Groups: Teleconsultation

SUMMARY:
The purpose is to evaluate the effectiveness and safety profile of telemedicine consultation system in making decision on IV thrombolysis.

DETAILED DESCRIPTION:
The rate of intravenous thrombolysis with tissue-type plasminogen activator or urokinase for stroke patients was extremely low in China. It has been demonstrated that telestroke may help to increase the rate of intravenous thrombolysis and improve the stroke care quality in the local hospitals. The aim of this study is to evaluate the effectiveness and safety of decision making of intravenous thrombolysis via telemedicine consultation system for acute ischemic stroke patients in China This trial network consists of one hub hospital (Xijing Hospital) and 14 spoke hospitals in the remote area of Shanxi Province. The telemedicine consultation system is an interactive, 2-way, wireless, audiovisual system based on portable hardwares--tablet computer or smartphone. Before this study, we have been investigating the usual stroke care quality in the spoke hospitals without the guidance from the hub hospital, which will be used as the historical control of this study. After that, the teleconsultation system will be introduced.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years and less than 80 years
* Acute ischemic stroke
* Presenting to Emergency Department of spoke hospitals within 4.5 hours of stroke symptom onset
* National Institutes of Health Stroke Scale (NIHSS) between 4 and 25
* Signed consent form by the patient or his relatives

Exclusion Criteria:

* Time of symptom onset unclear
* Unlikely to complete study through 3-month follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke patients arriving in the local hospitals within 4.5 hours of symptom onset
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients treated with intravenous thrombolysis | at 4.5 hours

SECONDARY OUTCOMES:
Favorite outcome at 3 months (modified Rankin score ≤2) | at 1 month/3 months
Stroke complications | at 24 hours/7days
  They include symptomatic intracranial hemorrhage (sICH), symptomatic cerebral edema from an original brain infarction, cerebral hernia, seizure, severe extracranial bleeding, pulmonary embolism, pulmonary edema, deep venous thrombosis, and sepsis.
Fatal and nonfatal cardiovascular events | at 7 days
  They include recurrent ischemic stroke, intracranial hemorrhage, subarachnoid hemorrhage, transient ischemic attack, myocardial infarction, angina and heart failure
All cause mortality | at 3 months
Time intervals | at 24 hours
  Those from stroke onset to arriving in emergency department(ED), and from arriving in ED to physician/CT initiation/CT interpretation/specific treatment.
Length of hospitalization | at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhirong Liu, MD, Principal Investigator — Xijing Hospital; Gang Zhao, MD, Study Director — Xijing Hospital
Locations (4):
- China (4):
  - Xingyuan Hospital, Yulin, Shanxi
  - Yulin First People's Hospital, Yulin, Shanxi
  - Yulin Second People's Hospital, Yulin, Shanxi
  - Yuyang District People's Hospital, Yulin, Shanxi

REFERENCES:
- [Derived] Yuan Z, Wang B, Li F, Wang J, Zhi J, Luo E, Liu Z, Zhao G. Intravenous thrombolysis guided by a telemedicine consultation system for acute ischaemic stroke patients in China: the protocol of a multicentre historically controlled study. BMJ Open. 2015 May 15;5(5):e006704. doi: 10.1136/bmjopen-2014-006704. PMID 25979867